CLINICAL TRIAL: NCT05276843
Title: Efficacy of Selected Exercises on Bone Mineral Density in Post-burn Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eman Mohamed othman (Other)
Responsible Party: Sponsor-Investigator, Eman Mohamed othman, professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00000000
Record Dates: First submitted 2022-02-28; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): receive Qigong exercise in addition to traditional physical therapy program
  Interventions: Combination Product: Qigong exercise program
- group B (No Intervention): receive traditional physical therapy program only

INTERVENTIONS:
Combination Product: Qigong exercise program — Qigong is a low-impact, weight-bearing exercise characterized by gentle movements designed to dissipate force throughout the body while the subject changes poses, with well-coordinated sequences of both isometric and isotonic segmental movements in the trunk and 4 extremities.
  Arms: group A

SUMMARY:
PURPOSE: to assess the efficacy of Qigong exercise on bone mineral density in post-burned patient.

BACKGROUND: During severe burns, more than 7% of the vertebral bone mineral density (BMD) is lost within 3-6 weeks of the injury and about 3% of the total body bone content is lost during the first 6 months after the injury.

Qigong exercise has been shown to be effective at attenuating declines in BMD and improving both balance performance and balance confidence in healthy middle-aged and older adults.

There are lack in knowledge and information in published studies about the efficacy of Qigong exercise on bone mineral density in post-burned patient.

So, this study will be designed to provide a guideline about the efficacy of Qigong exercise on bone mineral density in post-burned patient.

HYPOTHESES:

It will be hypothesized that:

It was hypothesized that Qigong exercise has no or limited effect in bone mineral density in post-burned patient.

RESEARCH QUESTION: Does Qigong exercise an effect on bone mineral density in post-burned patient?

DETAILED DESCRIPTION:
1. Measurement procedure:

   Bone density measurement was conducted before the first session and after two months of treatment.

   The test worked by measuring a specific bone or bones, usually the spine, hip and wrist. The density of these bones was then compared with an average index based on age, sex and size. The resulting comparison is used to determine risk for fractures and the stage of osteoporosis in an individual.

   Average bone mineral density = BMC/W (g/cm²).
   * BMC = bone mineral content = g/cm.
   * W = width at the scanned line. Data was graded according to Z score.

   Z-score:

   The Z-score is the comparison to the age matched normal subject. This is the number of standard deviations a patient's bone mineral density (BMD) differs from the average BMD of their age, sex and ethnicity. This value is used in premenopausal women, men under the age of 50, and in children. It is most useful when the score is less than 2 standard deviations below this normal. In this setting, it is helpful to scrutinize for coexisting illnesses that may contribute to osteoporosis such as glucocorticoid therapy, hyperparathyroidism or alcoholism. Z-score minus 1.5 and lower is considered below expected range of age, while Z-score above minus 1.5 is considered within expected range of age
2. Treatment procedures:

In this study the treatment protocol was presented in the form of an exercise program lasted for 50 minutes, twice weekly for 12 weeks postburn and consisted of weight bearing, strengthening and aerobic exercises and achieved under the following phases:

1. Warming up phase:

   The main aim of this phase was to get the muscles warm and loose for strength training. The subject has to train for ten minutes on a stationary bicycle at a mild velocity before the beginning of each exercise session. Bicycling helps direct needed blood flow to the muscles and prepares the body for exercise. Warming up is important for preventing injury as well as gaining maximal benefit from the exercise, because loose and warm muscles respond better to the challenge of the program.
2. Exercise phase:

Qigong is a low-impact, weight-bearing exercise characterized by gentle movements designed to dissipate force throughout the body while the subject changes poses, with well-coordinated sequences of both isometric and isotonic segmental movements in the trunk and 4 extremities. This style emphasizes slow and smooth movement involving major muscle groups, at a constant speed while practicing. The sway of its moment is usually centered, which makes it more safe for the elderly to practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients were 25-50 years old
* had thermal burn injuries of 2nd-3rd degree extended from the lower area of trunk to the lower extremities.
* the affected total body surface area of 30-45%.
* In the early burn stage (30-45 days in burn units), all patients were subjected to a unified physical therapy program consisted of positioning, range of motion, and gentle stretching exercises.

Exclusion Criteria:

* any history of endocrine, metabolic or other systemic diseases
* prior or ongoing supplementation with calcium
* previous or current bone-specific drugs or diseases affecting bone metabolism
* smoking
* any neurogenic disorder impairing sensory or motor function
* use of drugs known to affect the central nervous system or equilibrium
* previous brain injury or any disease affecting balance
* history of epilepsy
* previous or habitual high-intensity exercise
* lower extremity arthralgia
* lower extremity implant
* recent surgeries for heart or spine
* cancer
* hernia
* acute thrombosis
* kidney or bladder stones
* diabetes
* serious cardiovascular or cerebrovascular disease.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Bone density measurement | change in bone mineral density calculated at 8 weeks post treatment minus baseline.
  The test worked by measuring a specific bone or bones, usually the spine, hip and wrist. The density of these bones was then compared with an average index based on age, sex and size. The resulting comparison is used to determine risk for fractures and the stage of osteoporosis in an individual.

CONTACTS AND LOCATIONS:
Overall Officials: eman othman, PhD, Study Chair — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in bee venom or ulcer . we will share the results of this study within 1 year following publication.
Supporting Information: SAP, ICF
Time Frame: 1 year after publication
Access Criteria: the criteria will be assessed by the publication of the trial in an international journals.